CLINICAL TRIAL: NCT07048522
Title: Perioperative Nimodipine for Intra- and Postoperative Pain Management and Reduction of Anesthetic Requirements in Patients Undergoing Open Colectomy: a Prospective, Double-blind, Randomized Controlled Trial
Brief Title: Perioperative Intravenous Nimodipine Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Petros Tzimas, Professor of Anesthesiology, University of Ioannina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-4_2024-12-05
Record Dates: First submitted 2025-06-20; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Colectomy; Open Surgery; Pain; Pain, Postoperative; Pain, Acute
MeSH Terms: conditions — Pain; Pain, Postoperative; Acute Pain | interventions — Nimodipine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Forty patients (20 in each arm) undergoing surgical treatment for high-risk general surgery (open colectomy) will be included in this prospective, randomized, double-blind, controlled trial with two investigation arms: intervention arm (nimodipine). control arm (isotonic saline).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization and study medication will be handled by the hospital pharmacy. All research team members, caregiving clinicians and enrolled patients will be blinded to the study allocation arms and the randomization list will be concealed until all statistical analyses are made.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nimodipine (Experimental): Prepared (coded) by the pharmacy 50 ml solutions of nimodipine (2 mg/10 ml) with blinded 50 ml syringes will be used in each patient.
  Interventions: Drug: Nimodipine
- Isotonic saline (Placebo Comparator): Prepared (coded) by the pharmacy 50 ml solutions with blinded 50 ml syringes of isotonic saline will be used in each patient.
  Interventions: Drug: Isotonic Saline

INTERVENTIONS:
Drug: Nimodipine — A continuous dose of 4 mg/h (20 ml/h) of nimodipine solution will be administered continuously 1 h prior to start of operation until 1 h after start of the procedure. • The nimodipine dose will be then reduced to 2 mg/h (10 ml/h) until 24 hrs after the end of the procedure.
  Arms: Nimodipine
Drug: Isotonic Saline — A continuous dose of 20 ml/h of normal saline solution will be administered continuously one (1) h prior to start of operation until 1 h after start of the procedure. The normal saline dose will be then reduced to 10 ml/h until 24 h after the end of the procedure.
  Arms: Isotonic saline

SUMMARY:
The role of perioperative IV administration of nimodipine, an L-type calcium channel antagonist which is capable of crossing the blood-brain barrier, on peri-operative opioid and anesthetics requirements, pain intensity, opioid-related side effects and early postoperative bowel mobility in patients undergoing surgical treatment for bowel cancer with open radical colectomy remains scarcely explored. A prospective double-blind, randomized controlled trial investigating the effect of perioperative IV administration of nimodipine in patients undergoing open colectomy for cancer treatment is therefore conducted.

DETAILED DESCRIPTION:
Background with aim: Acute postoperative pain is still of major clinical concern for a large number of patients undergoing surgery worldwide. Despite advances in pain management strategies, many patients continue to suffer from moderate-to-severe pain during the early postoperative period, while opioids are still largely over-prescribed. Not effectively and especially unrelieved pain can result in decreased patient satisfaction, increased morbidity, prolonged hospital length-of-stay and increased risk of persistent pain. Furthermore, effective treatment of acute postoperative pain using opioid analgesics remains the core treatment for postoperative pain. Although the potential benefits of opioid therapy for acute pain lead to a short-term pain control there are several potential severe side-effects associated with opioid use which may outweigh the benefits including sedation, nausea, vomiting, constipation especially in bowel surgery, and the risk of long-term use. Although various non-opioid drugs have been investigated over the past decades, information regarding L-type calcium channel blockers in acute postoperative pain is limited. In this respect, the perioperative use of nimodipine, a drug which furthermore crosses the blood-brain barrier and has direct effects on the Central Nernous System (CNS) could potentiate the effects of opioid analgesia and intraoperative anesthetic requirements, providing improved analgesia and potentially reduce for opioids in the perioperative period. Therefore, the investigators decided to carry out the present study with the aim to examine the analgesic efficacy and safety of perioperatively administered IV nimodipine in patients undergoing open colectomy on perioperative opioid and anesthetic consumption, pain intensity, opioid-related side effects and early postoperative bowel mobility.

Method: A power analysis based on a previous preliminary study using IV nimodipine for medium risk general surgery (open cholecystectomy) showed that 9 patients would provide a power greater than 0.9 (α = 0.05) for detection of differences of pain scores and cumulative opioid consumption over time (up to 48 h). Therefore, 40 patients undergoing open colectomy will be included in this prospective, randomized, double-blind, controlled trial with two arms: an intervention arm (IV nimodipine 4 mg/h starting 1h prior to surgery until one h after the start of surgery, followed by 2 mg/h until 24 h post-operation) and a control arm (isotonic saline 20 ml/ h 1h prior to and until one h after start of surgery, followed by 10 ml/h until 24 h post-operation). The study is approved by the local hospital scientific board (#18-4_2024-12-05).

Hypothesis: The investigators hypothesize that perioperative intravenous administration of nimodipine, an L-type calcium channel antagonist, will be effective in reducing intraoperative anesthetic requirements, as well as intra- and postoperative opioid requirements, as well as postoperative pain intensity and opioid-related side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for open surgical treatment of bowel cancer at the General Hospital of Patra

Exclusion Criteria:

* Age < 18 years, > 75 years
* American Society of Anesthesiologists (ASA) physical status > III
* Allergy to nimodipine
* Inability to provide informed consent
* Known severe renal insufficiency
* Known severe bradyarrhythmia
* Daily opioid consumption the last 7 days before surgery
* Pain intensity assessed using the Numerical Rating Scale (NRS; 0-10), with scores greater than 5 reported on more than half of the days during the past month.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-05-19 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Intraoperative Remifentanil Consumption | Intraoperative period, defined as the time (in minutes) from induction of general anesthesia to extubation.
  Remifentanil will be administered intraoperatively based on qNOX (quantum NOXious stimulus index) levels, which will be maintained between 40 and 60. qNOX values below 40 will prompt a reduction in remifentanil dosing, while values above 60 will prompt an increase, in order to optimize analgesia.
Intraoperative propofol consumption | Intraoperative period, defined as the time (in minutes) from induction of general anesthesia to extubation.
  Propofol will be administered intraoperatively based on BIS (Bispectral Index) and qCON (quantum Consciousness Index) values, which will be maintained between 40 and 60. BIS or qCON values below 40 will prompt a reduction in propofol dosing, while values above 60 will prompt an increase, in order to maintain appropriate depth of anesthesia.
Cumulative opioid consumption within 0 to 72 hours postoperatively | From Post Anesthesia Care Unit (PACU) admission (time zero) to 72 hours postoperatively.
  Cumulative morphine consumption (mg) during the first 72 hours after arrival at the Post Anesthesia Care Unit (PACU). During the first hour in the PACU, morphine will be administered using a titration method. Following transfer to the surgical ward, a patient-controlled analgesia (PCA) device will be used to monitor morphine consumption. Cumulative opioid use will be recorded at specific time points: 3, 6, 12, 18, 24, 30, 36, 48, 60, and 72 hours postoperatively.

SECONDARY OUTCOMES:
Pain intensity at rest | From Post Anesthesia Care Unit (PACU) admission (time zero) to 72 hours postoperatively.
  Pain intensity at rest will be assessed using the Numerical Rating Scale (NRS; 0-10), starting upon arrival at the Post Anesthesia Care Unit (PACU) and continuing at the following postoperative time points on the ward: 3, 6, 12, 18, 24, 30, 36, 48, 60, and 72 hours.
Pain intensity during coughing | From Post Anesthesia Care Unit (PACU) admission (time zero) to 72 hours postoperatively.
  Pain intensity during coughing will be assessed using the Numerical Rating Scale (NRS; 0-10), beginning upon arrival at the Post Anesthesia Care Unit (PACU) and at the following postoperative time points on the ward: 3, 6, 12, 18, 24, 30, 36, 48, 60, and 72 hours.
Opioid related sedation | From Post Anesthesia Care Unit (PACU) admission (time zero) to 72 hours postoperatively.
  Number of participants with postoperative sedation assessed using the Ramsay Sedation Scale (range: 1 = anxious/agitated to 6 = no response to stimulus).
Opioid related pruritus | From Post Anesthesia Care Unit (PACU) admission (time zero) to 72 hours postoperatively.
  Number of participants with documented pruritus related to opioid use, recorded as a binary outcome variable (yes/no).
Postoperative nausea and/or vomiting (PONV) | From Post Anesthesia Care Unit (PACU) admission (time zero) to 72 hours postoperatively.
  Number of participants with documented postoperative episodes of nausea and/or vomiting, recorded as a binary outcome variable (yes/no).
Time to first signs of bowel mobilization | From end of surgery to 90 hours postoperatively or until hospital discharge, whichever comes first.
  Time (in hours) from the end of surgery to the first documented sign of bowel function, defined as either the first bowel sounds on auscultation or the first passage of flatus. Assessment will take place in the surgical ward at the following postoperative time points: 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, and 90 hours, or until hospital discharge, whichever comes first.
Length of stay (LOS) | Duration of hospitalization, from the day of admission to the day of discharge (up to 30 days).
  Total duration of hospitalization, measured in days from admission to discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Petros Tzimas, MD, PhD, Principal Investigator — University of Ioannina, Greece
Locations (1):
- St. Andrews General Hospital of Patras, GREECE, Pátrai, Achaea, Greece

IPD SHARING:
Plan to Share IPD: No
The data will be shared upon reasonable request by other researchers